CLINICAL TRIAL: NCT05909137
Title: Feasibility of Omitting Clinical Target Volume in Radical Treatment of Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: Omitting Clinical Target Volume in Radical Treatment of Unresectable Stage III Non-small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director of oncology department，clinical professor, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-022
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Immunotherapy; Intensity Modulated Radiation Therapy; Radiotherapy; NSCLC
Keywords: IMRT; immunotherapy; CTV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: CTV-omitted IMRT+adjuvant immunotherapy
  Interventions: Radiation: IMRT+adjuvant immunotherapy
- control group: CTV-delineated IMRT+adjuvant immunotherapy
  Interventions: Radiation: IMRT+adjuvant immunotherapy

INTERVENTIONS:
Radiation: IMRT+adjuvant immunotherapy — The enrollment was randomly (1:1) assigned into the study group with CTV-omitted IMRT and the control group with CTV-delineated IMRT using a random number table.

SUMMARY:
Simultaneous radiotherapy followed by adjuvant immunotherapy is the standard treatment modality of unresectable stage III NSCLC. Our preliminary study confirmed that the treatment of CTV-omitted IMRT regimen did not compromise the PFS or OS and significantly reduced the incidence of severe radiation pneumonia and radiation esophagitis.

The purpose of this study was to observe the role of radiotherapy modalities that omit CTV in the context of immunotherapy for NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* •Patients with advanced (Stage IIIA or IIIB AJCC 7) NSCLC that was histologically or cytologically inoperable

  * ECOG whole body status (performancestatus,PS) level 0 or 1
  * The estimated survival time is more than 12 weeks, 18 ~80 years old
  * Laboratory results within 2 weeks prior to radiotherapy met the following criteria: ① Neutrophil count > 1,500/ MCL Heathko-Pilot Oncology Research Fund; ② Platelet > 50,000/ MCL; ③ Total bilirubin < 1.5 times of the normal upper limit value; ④AST(SGOT)/ALT(SGPT) < 2.5 times of the normal upper limit; ⑤ Serum creatinine < 1.5 times of the normal upper limit value; ⑥ The results of coagulation function examination were within the normal range
  * Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy tests (serum or urine) within 7 days before admission, and the results are negative, and are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the trial drug. For men, they must agree to use appropriate methods of contraception or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug
  * Understand and voluntarily sign written informed consent
  * The investigator judged that the patient had good compliance

Exclusion Criteria:

* Malignant pleural/pericardial effusions, previous thoracic radiotherapy or chemotherapy
* Uncontrolled concurrent diseases, including but not limited to symptomatic congestive heart failure, unstable angina pectoris and myocardial infarction, uncontrolled grade III hypertension, liver insufficiency, renal insufficiency, uncontrolled diabetic blood sugar, arrhythmia, mental illness or social condition, etc.
* Pregnant or nursing women
* The patient has no history of intracranial hemorrhage or spinal cord hemorrhage
* HIV-positive patients receiving combination antiretroviral therapy
* Active tuberculosis
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Prior allogeneic stem cell or solid organ transplantation
* Researchers determine other conditions that may affect the conduct of clinical studies and the determination of their findings

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with advanced (Stage IIIa or IIIb) NSCLC that was histologically or cytologically inoperable.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | through study completion，up to 12 weeks
  The time between randomization and the first occurrence of disease progression or die
radiation respiratory events or esophagitis with grade 3 or higher | after radiation therapy，up to 1 year

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 year
  Time from randomization to death from any cause

IPD SHARING:
Plan to Share IPD: No